CLINICAL TRIAL: NCT03273647
Title: Adjuvant Radiotherapy for T3N0M0 Esophageal Squamous Cell Carcinoma With Positive Circumstantial Resection Margin(a Randomized Controlled Trial)
Brief Title: Adjuvant Radiotherapy for Esophageal Squamous Cell Carcinoma With Positive Circumstantial Resection Margin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jiaqing Xiang, Professor of Department of Thoracic Surgery, Fudan University Shanghai Cancer Center, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO-CRM
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Esophageal Squamous Cell Carcinoma; Positive Circumferential Resection Margin
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgery plus radiation (Experimental): adjuvant radiotherapy is developed in this arm
  Interventions: Radiation: radiation
- surgery alone (No Intervention): No adjuvant radiotherapy,that is surgery alone is developed in this arm

INTERVENTIONS:
Radiation: radiation — A total dose of 40Gy will be delivered in 20 fractions at 2.0Gy/fraction, 5 fractions per week in 4 weeks.
  The CTV encompassed the bilateral supraclavicular region, all mediastinal lymph nodes, the anastomosis site, and the left gastric and Celiac nodes.
  Arms: surgery plus radiation

SUMMARY:
The purpose of this study is to determine the efficacy of adjuvant radiotherapy for esophageal squamous cell carcinoma with positive circumstantial resection margin.

DETAILED DESCRIPTION:
Although preoperative chemoradiation therapy followed by surgery is the most common approach for patients with resectable esophageal cancer, the considerable number of esophageal cancer patients received operation as the first treatment modality. Accordingly, postoperative treatments have been playing an important role because of the poor survival rates of the patients who have been treated with resection alone. The existing data shows that the 5-yeal survival rate of stage T2-3N0M0(UICC 7th edition) of thoracic esophageal squamous cell carcinoma(TESCC) after surgery is about 50% ,and locoregional lymph nodes metastases is responsible for the main cause of failure while distal metastases account for relatively less ratio. Therefore, the subclinical residual tumor is affirmative even if the early disease has been undergone curable excision and local adjuvant treatment may be essential. In rectal cancer, the involvement of the circumferential resection margin (CRM) is one of the key factors for local recurrence and poor prognosis,based on reports in which CRM with < 1mm was found to be prognostically significant, whereas the clinical and prognostic significance of the CRM involvement in EC has been investigated only in a few series showing conflicting results, as some studies suggest a significant influence of CRM. There is lack of clear evidence for prophylactic radiation therapy in positive Circumferential Resection Margin(CRM) patients of TESCC now. In view of this, the randomized controlled trial will determine the clinical efficacy and toxicity of adjuvant radiotherapy in positive Circumferential Resection Margin(CRM) for thoracic esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Patients with esophageal cancer who received R0 operations in Fudan University Shanghai Cancer Center and postoperative pathology: squamous cell cancer,positive Circumferential Resection Margin(CRM)+

* KPS≥70 before radiotherapy;
* Did not receive neoadjuvant or adjuvant treatment;
* No clear recurrent or metastatic lesions before radiotherapy;
* Intensity modulated radiation therapy(IMRT) is accepted;
* Regular follow-up.

Exclusion Criteria:

* Exploratory thoracotomy or palliative surgery;
* No clear recurrent or metastatic sites;
* Recurrence or metastasis is not certain;
* death of no definite cause.
* Irregular follow-up;

Ages: 18 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival time | up to 3 years
  including survival time from randomization to locoregional recurrence and to distal metastasis

SECONDARY OUTCOMES:
overall survival time | up to 3 years
  survival time from randomization to death

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqing Xiang, MD, Principal Investigator — professor of Department of Thoracic Surgery, Fudan University Shanghai Cancer Center

IPD SHARING:
Plan to Share IPD: No